CLINICAL TRIAL: NCT02200575
Title: Pharmacovigilance and Patient Compliance in Hypertensive Patients. Observational Study
Brief Title: Pharmacovigilance and Patient Compliance in Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.359
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with non-secondary, essential hypertension
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®

SUMMARY:
Study to confirm the safety profile of telmisartan (benefit-risk ratio) under normal conditions of use after market launch and to supplement the present data on the safety of telmisartan. Furthermore to assess effectiveness of a single dose of telmisartan per day to control blood pressure for 24 hours, especially during the last few hours of the dosage interval. Additionally to evaluate compliance with treatment, as an indirect measurement, and to confirm the efficacy and possible risks associated with treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients of either sex over the age of 18 years suffering from non-secondary essential hypertension with values of at least 90 mmHg (diastolic) and 140 mmHg (systolic)

Exclusion Criteria:

- corresponding to the contraindications listed in the summary of product characteristics of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients over 18 years of age suffering non-secondary, essential hypertension, treated by general practitioners and/or specialists
Sampling Method: Non-Probability Sample
Enrollment: 10333 (Actual)
Dates: Start 1999-05; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in heart rate | Baseline, up to 8 weeks after start of treatment
Assessment for patients with changes in laboratory values | Baseline, up to 8 weeks after start of treatment
Number of patients with adverse events | Up to 8 weeks after start of treatment

SECONDARY OUTCOMES:
Changes in mean systolic and diastolic blood pressure values | Baseline, up to 8 weeks after start of treatment
  Measured by means of ambulatory blood pressure monitoring (ABPM) over 24 hours
Changes in mean systolic and diastolic blood pressure values | Baseline, up to 8 weeks after start of treatment
  Measured three times at intervals of two minutes with the patient seated and lying down for 5 minutes, using a sphygmomanometer
Evaluation of treatment compliance as percentage of tablets planned | Up to 8 weeks after start of treatment
  (number of tablets taken / total number of days) x 100